CLINICAL TRIAL: NCT02559362
Title: Study on Breast Cancer Patient Perspectives of Exercise
Status: Completed | Type: Observational
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: UPCC 23114
Record Dates: First submitted 2015-06-19; First posted 2015-09-24 (Estimated); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Survey

SUMMARY:
The goal of the study is to establish the feasibility/willingness of breast cancer patients to delay surgery to do an exercise program, or be randomized to an exercise training program following treatment, and to see if that willingness correlates with prior physical activity history.

ELIGIBILITY:
Inclusion Criteria:

* women,
* breast cancer diagnosis,
* all races will be included.

Exclusion Criteria:

* men,
* those with no breast cancer (ductal carcinoma in situ),
* pregnant women,
* children

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast cancer subjects
Sampling Method: Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-06-03 (Actual)

PRIMARY OUTCOMES:
Number of subjects providing completed surveys | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Schmitz, PhD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States